CLINICAL TRIAL: NCT04695405
Title: Genetic Markers Associated With Response to Intravenous Ketamine
Brief Title: Pharmacogenetics Associated With IV Ketamine
Status: Completed | Type: Observational
Sponsor: Brain and Cognition Discovery Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: Ket-PGx
Record Dates: First submitted 2020-12-28; First posted 2021-01-05 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients will provide two saliva samples containing genetic information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment-Resistant Depression: Patients, who previously received intravenous ketamine, will be asked to provide genetic samples in order to assess relationships between response and genetic markers.
  Interventions: Genetic: Saliva Genetic Samples

INTERVENTIONS:
Genetic: Saliva Genetic Samples — Patients will provide two saliva swabs containing genetic materials.

SUMMARY:
The Canadian Rapid Treatment Center of Excellence (CRTCE) is a healthcare facility principally focused on providing best practices of intravenous ketamine treatment to adult patients suffering from treatment resistant depression. Patients who have received IV ketamine at the clinic are eligible to participate in this study where genetic biomarkers are correlated with response to IV ketamine.

ELIGIBILITY:
Inclusion Criteria:

1. Must have received IV ketamine previously to treat Treatment-Resistant Depression
2. Between the ages of 18-65 years old.
3. Clinical diagnosis of MDD
4. Individuals may have had comorbid psychiatric conditions (e.g., anxiety), but the comorbid psychiatric condition cannot be the primary clinical concern.
5. Ability to provide informed consent

Exclusion Criteria:

1. Individuals who meet DSM 5 criteria for a substance use and/or alcohol use disorder in the past 3 months.
2. Individuals who are currently experiencing psychotic symptoms as part of an MDE (mood congruent/mood incongruent).
3. Individuals who are unable to consent to the procedure.
4. Individuals who are unable to adhere to the protocol in its totality

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants will have received IV ketamine previously for treatment resistant depression, as defined by the DSM-5
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
Genetic Biomarkers | 1 month
  Genetic markers associated with metabolism of IV ketamine will be assessed
Quick Inventory of Depressive Symptomatology Self Report 16-Item | Over 1-2 weeks
  The QIDS-SR16 is a self-report assessment used to evaluate depression severity in patients with a Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, diagnosis of Major Depressive Episode. In total, there are 16 individual questions evaluating 9 DSM domains. The highest score is 27, indicating severe depression, while the lowest score is 0, which would suggest a complete absence of depressive symptoms.
Generalized Anxiety Disorder 7-item | Over 1-2 weeks
  The GAD-7 is a 7 item self-report assessment used to evaluate symptoms of anxiety. The scale ranges from 0 (not at all) to 3 (nearly every day). To total score ranges from 0 suggesting a lack anxiety symptoms to 21, indicating severe anxiety.
Snaith-Hamilton Pleasure Scale | Over 1-2 weeks
  The SHAPS assessment is a 14 item self report tool used to measure anhedonia. Each item can be have a response of 1 (Definitely agree), 2(Agree), 3(Disagree), and 4(definitely disagree). The total score ranges from 14 to 56, in which higher scores on the assessment indicate higher levels of anhedonia.
Sheehan Disability Scale | Over 4 initial infusions
  The SDS contains 3 items, each ranging between zero to ten. The SDS is a self-reported assessment of disability within the context of depression. The total score ranges from 0, indicating no impairment, to 30, indicating severe impairment.
Clinician Administered Dissociative States Scale | Over 1-2 weeks
  The CADSS is a 23-item assessment administered by a clinician in order to evaluate dissociative symptoms. Each item is evaluated on a scale from 0, suggesting no dissociative symptom, to 4, suggesting extreme dissociation. In total, patients can score between 0 to 92, indicating extreme dissociation.

SECONDARY OUTCOMES:
Work Productivity and Activity Impairment Questionnaire (WPAI) | 1 month
  WPAI is a questionnaire used to evaluate lost productivity due to depression. scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity.
Mystical Experience Questionnaire (MEQ) | 1 month
  Mystical Experience Questionnaire (MEQ) is a self-report measure that has been used to assess the effects of hallucinogens in laboratory studies. Some studies suggest that mysticism may be associated with a response to ketamine. The MEQ is a 30 item questionnaire, with each item ranging from 0 to 5. A higher score denotes a strong mystical experience.
Childhood Trauma Questionnaire (CTQ) | 1 month
  The CTQ assesses five types of childhood trauma: 1)Emotional neglect 2) physical abuse 3) emotional abuse 4)physical neglect 5) sexual abuse.
  Each item being rated in 5 answer choice from 1 to 5 (never, rarely, sometimes, often or very often)
UCLA Loneliness Scale (UCLA) | 1 month
  20 item Self report scale measuring loneliness. Scales range from 0 to 60 with higher scores indicating a higher level of loneliness.
Diet Screener Questionnaire | 1 month
  Captures data regarding an individuals dietary habits over the past month
Quality of Life Questionnaire (EQ-3D-5L) | 1 month
  EQ-5D-5L measures health outcome self-completed by respondents. It consists of EQ-5D-5L descriptive system and EQ visual analogue scale (EQ-VAS). The descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each has 5 levels (1-no problem, 2-slight problems, 3-moderate problems, 4-severe problems, 5-extreme problems). The responses are used to generate Health Status Index (HSI). HSI range is -0.148 to 0.949, is anchored at 0 (dead) and 1 (full health).
Perceived Health Questionnaire (PHQ) | 1 month
  PHQ-9 is 9-item, self-reported scale assessing 9 symptom domains of Diagnostic and Statistical Manual of Mental Disorders, Major Depressive Disorder criteria. Each item is rated on 4-point scale (0 = Not at all, 1 = Several Days, 2 = More than half days, 3 = Nearly every day). The scores are summed for a total score ranging from 0-27. Higher score indicates greater severity of depression. Severity of PHQ-9 categorized as follows: None-minimal (0-4), Mild (5-9), Moderate (10-14), Moderately Severe (15-19), Severe (20-27). The recall period is 2 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua D Rosenblat, MD, MSc, Principal Investigator — Canadian Rapid Treatment Center of Excellence
Locations (1):
- Canadian Rapid Treatment Centre of Excellence, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to confidentiality. Only aggregate data will be published or made available.